CLINICAL TRIAL: NCT01175798
Title: Immunologic Impact of Vitamin D Repletion in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Impact of Vitamin D Repletion in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehrotra, Anita, M.D. (Individual)
Collaborators: National Kidney Foundation, United States (Other); American Heart Association (Other)
Responsible Party: Principal Investigator, Anita Mehrotra MD, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-2275
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Vitamin D Deficiency; End-stage Renal Disease
Keywords: Vitamin D deficiency; End-stage renal disease; Immunity
MeSH Terms: conditions — Vitamin D Deficiency; Kidney Failure, Chronic | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No treatment (standard of care) (No Intervention): Patients will be randomized in a 3:2 ratio to oral Vitamin D treatment, or standard of care (no repletion).
- Vitamin D repletion (Experimental): Patients will be randomized in a 3:2 ratio to oral Vitamin D treatment, or standard of care (no repletion).
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 50,000 IU PO weekly x 6 weeks
  Other Names: Vitamin D
  Arms: Vitamin D repletion

SUMMARY:
Dialysis patients often suffer from defects in their immune system (that part of the body which fights infection). Evidence suggests that Vitamin D deficiency may have a negative effect on immunity, and many dialysis patients are deficient in Vitamin D. We believe that by giving Vitamin D to dialysis patients who are deficient, we may help improve their immune system. This study will test that idea.

DETAILED DESCRIPTION:
Innate and adaptive immunity are commonly impaired in patients with end stage renal disease (ESRD) on dialysis. The myriad of immune defects in these patients, often attributed to uremia, may account for their high risk of bacterial infection and suboptimal responses to vaccination. The mechanisms underlying these abnormalities in immune function remain elusive, but emerging evidence indicates that 25OH-Vitamin D exerts potent and complex control over innate and adaptive immunity. Vitamin D deficiency is common in dialysis patients, and the immune effects associated with 25OH-Vit D deficiency overlap with those found in many dialysis patients. The kidney is the dominant site of 1-alpha-hydroxylase activity required for producing active 1,25OH-Vit D; however, immune cells also express the 1-alpha-hydroxylase enzyme. Evidence indicates the effects of Vitamin D on modulating immunity require conversion of 25OH-Vit D to 1,25OH-Vit D within the immune cells (rather than via circulating 1,25OH-Vit D). As a consequence, total body deficiency of 25OH-Vit D can impact immune function despite ongoing therapy with active 1,25OH-Vit D (which most dialysis patients are receiving). Our preliminary data confirm the high prevalence of 25OH-Vit D deficiency in dialysis patients and show that Th1 T cell alloimmunity is stronger in patients deficient in 25OH-Vit D, supporting the hypothesis that Vit D deficiency has important immunological consequences. Based on the published literature and our preliminary data, we hypothesize that repletion of 25OH-Vit D enhances immunity in dialysis patients. To test this hypothesis, we propose a randomized controlled trial of oral 25OH-Vit D repletion in this patient population. One hundred fifty 25OH-Vit D deficient study subjects will be randomized to either treatment with 50,000 IU oral 25OH-Vit D weekly or no treatment (standard of care). The primary outcome of change in 25OH-Vit D level will be measured at 6 weeks, 3 months, 6 months, and 12 months. Secondary outcomes to be measured include change in peripheral blood mononuclear cell (PBMC) profile by flow cytometry at 6 and 12 months, change in ELISPOT-based panel of reactive T cell (PRT) readout at 6 and 12 months, change in PMBC cytokine production in response to toll-like-receptor stimulation at 6 and 12 months, and response to influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Chronic hemodialysis treatments for at least 2 consecutive months
3. 25OH-Vitamin D level < 25 ng/mL (inclusion criteria for randomization)

Exclusion Criteria:

1. History of acute renal failure requiring dialysis with potential for renal recovery
2. History of HIV/AIDS
3. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Mehrotra, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Li L, Lin M, Krassilnikova M, Ostrow K, Bader A, Radbill B, Uribarri J, Tokita J, Leisman S, Lapsia V, Albrecht RA, Garcia-Sastre A, Branch AD, Heeger PS, Mehrotra A. Effect of cholecalciferol supplementation on inflammation and cellular alloimmunity in hemodialysis patients: data from a randomized controlled pilot trial. PLoS One. 2014 Oct 8;9(10):e109998. doi: 10.1371/journal.pone.0109998. eCollection 2014. PMID 25296334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Treatment (Standard of Care) | Vitamin D Repletion
Started | 34 | 62
Completed | 27 | 41
Not Completed | 7 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment (Standard of Care) | Vitamin D Repletion | Total
Number analyzed (Participants) | 34 | 62 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (14.9) | 60.2 (14.3) | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 26 | 40
  Male | 20 | 36 | 56
25(OH) vitamin D [Median (Inter-Quartile Range); unit: ng/dL] | 13.1 [9.9 to 18.6] | 13.4 [9.3 to 19.7] | 13.2 [9.5 to 19.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in 25OH-Vitamin D Level
Description: Vitamin D deficient study subjects will be randomized to either treatment with 50,000 IU oral 25OH-Vit D weekly or no treatment (standard of care). The primary outcome of change in 25OH-Vit D level will be measured at 6 weeks, 3 months, 6 months, and 12 months.
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | No Treatment (Standard of Care) | Vitamin D Repletion
Number analyzed (Participants) | 27 | 41
ng/dL | 15.8 [9.5 to 19.5] | 40.9 [32.2 to 45.5]

2. Secondary Outcome: Change in Immune Parameters
Description: Secondary outcomes to be measured include change in peripheral blood mononuclear cell (PBMC) profile by flow cytometry at 6 and 12 months, change in ELISPOT-based panel of reactive T cell (PRT) readout at 6 and 12 months, change in PMBC cytokine production in response to toll-like-receptor stimulation at 6 and 12 months, and response to influenza vaccination.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | No Treatment (Standard of Care) | Vitamin D Repletion
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/62
Other Adverse Events (participants affected / at risk) | 0/34 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes